CLINICAL TRIAL: NCT01084525
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 1B Study of OTO-104 Given as a Single Intratympanic Injection in Subjects With Unilateral Meniere's Disease
Brief Title: OTO-104 for Meniere's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Carl LeBel, PhD, Chief Scientific Officer, Otonomy, Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 104-200901
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Meniere's Disease
Keywords: Meniere's Disease; Vertigo; Definitive vertigo; Vertigo episodes; Vertigo frequency; Tinnitus; Hearing loss; Aural Fullness
MeSH Terms: conditions — Meniere Disease; Vertigo; Tinnitus; Hearing Loss | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- OTO-104 (steroid) 3 mg (Experimental)
  Interventions: Drug: OTO-104 (steroid) 3 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- OTO-104 (steroid) 12 mg (Experimental): The start of 12 mg dose cohort is contingent on safety data from 3 mg dose cohort.
  Interventions: Drug: OTO-104 (steroid) 12 mg

INTERVENTIONS:
Drug: OTO-104 (steroid) 3 mg — OTO-104 3 mg dose cohort, single intratympanic injection.
  Arms: OTO-104 (steroid) 3 mg
Drug: Placebo — Placebo arm will be conducted in parallel with each OTO-104 dose cohort.
  Arms: Placebo
Drug: OTO-104 (steroid) 12 mg — Sequential dose cohort escalation to OTO-104 12 mg dose cohort will occur pending the safety evaluation of 28 day follow up safety data for the OTO-104 3 mg dose cohort. OTO-104 12mg dose cohort is also a single intratympanic injection.
  Arms: OTO-104 (steroid) 12 mg

SUMMARY:
The purpose of this study is to evaluate the safety of OTO-104 in subjects with unilateral Meniere's disease. The effectiveness of OTO-104 to reduce the symptoms of Meniere's disease will also be evaluated.

DETAILED DESCRIPTION:
Meniere's disease is a debilitating disorder of the inner ear which includes symptoms such as vertigo, tinnitus, hearing loss and aural fullness. Meniere's disease may result from an imbalance of fluid in the inner ear. Several studies have shown that corticosteroids may help manage this imbalance yet the effect does not last very long. OTO-104 is a longer lasting corticosteroid which could provide significant benefit to patients with Meniere's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a diagnosis of unilateral Meniere's disease by 1995 American Academy of Otolaryngology - Head and Neck Surgery (AAOHNS) criteria and reports active vertigo for the 2 months prior to the study lead-in period.
2. Subject has experienced active vertigo during the lead-in period.
3. Subject has asymmetric low frequency sensorineural hearing loss.
4. Subject agrees to maintain their current treatments for Meniere's disease while on-study.
5. Subjects not currently on a low-salt diet or diuretic should have a medical history of having used one or both of these treatments for at least 1 month without relief of symptoms.
6. Subjects currently on a low-salt diet and/or diuretic at the time of screening agree to continue this treatment throughout the study.

Exclusion Criteria:

1. Subject has an infection in the ear, sinuses, or upper respiratory system.
2. Subject is pregnant or lactating.
3. Subject has a history of immunodeficiency disease.
4. Subject has a history of previous endolymphatic sac surgery.
5. Subject has a history of previous use of intratympanic (IT) gentamicin in the affected ear.
6. Subject has a history of tympanostomy tubes with evidence of perforation or lack of closure.
7. Subject has experienced an adverse reaction to IT injection of steroids.
8. Subject has used an investigational drug or device in the 3 months prior to screening.
9. Subject has had a duration of Meniere's disease of >20 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the safety and tolerability of two ascending OTO-104 doses relative to placebo. Safety assessments will be performed for 3 months post single intratympanic injection of OTO-104 or placebo. | 3 months

SECONDARY OUTCOMES:
The secondary objective of this study is to evaluate the clinical activity of two OTO-104 doses relative to placebo. Change in baseline for vertigo frequency will be evaluated with descriptive statistics. | 3 months
The impact of tinnitus on activities of daily living will be measured. | 3 months
Hearing loss in the affected ear will be measured by audiometric examination. | 3 months
Quality of life will be measured by patient reported questionnaire. | 3 months
Severity of vertigo episodes will be measured by the patient reported vertigo score. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Chair — Otonomy, Inc.
Locations (15):
- United States (15):
  - House Ear Institute, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Colorado Otolaryngology Associates, Colorado Springs, Colorado
  - Silverstein Institute, Sarasota, Florida
  - Northwestern University, Feinberg School of Medicine, Otolaryngology, Chicago, Illinois
  - Mass Eye & Ear Infirmary, Boston, Massachusetts
  - University of Michigan Hospitals, Dept. of Otolaryngology, Ann Arbor, Michigan
  - Michigan Ear Institute, Farmington Hills, Michigan
  - St Louis University, St Louis, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Crescent Medical Research, Salisbury, North Carolina
  - Wilmington Medical Research, Wilmington, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University Of Texas, Southwestern Medical Center, Dallas, Texas